CLINICAL TRIAL: NCT03749187
Title: A Target Validation/Phase1 Study of BGB-290 in Combination With Temozolomide in Adolescent and Young Adult IDH1/2 Newly Diagnosed and Recurrent Mutant Gliomas
Brief Title: BGB-290 and Temozolomide in Treating Isocitrate Dehydrogenase (IDH)1/2-Mutant Grade I-IV Gliomas
Acronym: PNOC017
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: BeiGene USA, Inc. (Industry)
Responsible Party: Principal Investigator, Sabine Mueller, MD, PhD, Professor, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18083; NCI-2018-02345 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PNOC017 (Other: Pediatric Neuro-Oncology Consortium (PNOC))
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma; IDH1 Gene Mutation; IDH2 Gene Mutation; Low Grade Glioma; Malignant Glioma; Recurrent Glioblastoma; Recurrent WHO Grade II Glioma; Recurrent WHO Grade III Glioma; WHO Grade II Glioma; WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — pamiparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Pamiparib (BGB-290), Temozolomide (TMZ)) (Experimental): Participants with grades III-IV newly diagnosed IDH1/2 mutant glioma receive 60mg pamiparib (BGB-290) PO BID on days 1-28 and 20mg temozolomide (TMZ) PO daily on days 1-21. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide (TMZ)
- Arm B (BGB-290, Temozolomide) (Experimental): Participants with grades I-IV recurrent IDH1/2 mutant glioma receive 60mg PARP inhibitor pamiparib (BGB-290) PO BID on days 1-28 and 20mg temozolomide PO daily on days 1-21. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Cohort B0: Participants who are surgical candidates with grades I-IV recurrent IDH1/2 mutant glioma receive 60mg PARP inhibitor BGB-290 PO BID for 7 days, pre-surgery. After recovery from surgery, participants receive PARP inhibitor BGB-290 PO BID on days 1-28 and 20mg temozolomide PO daily on days 1-21. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: PARP Inhibitor BGB-290 — Given PO
  Other Names: BGB-290; Pamiparib
Drug: Temozolomide (TMZ) — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; temozolomide

SUMMARY:
This phase I trial studies the side effects and best dose of BGB-290 and temozolomide in treating adolescents and young adults with IDH1/2-mutant grade I-IV glioma that is newly diagnosed or has come back. BGB-290 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving BGB-290 and temozolomide may work better in treating adolescents and young adults with IDH1/2-mutant grade I-IV glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of the combination of Poly (ADP-Ribose) polymerase (PARP) inhibitor BGB-290 (BGB-290) and temozolomide (TMZ) in adolescent and young adult (AYA) subjects with IDH1/2-mutant glioma, including the maximum tolerated dose (MTD) and characterization of dose-limiting toxicities (DLTs) in both, newly diagnosed and recurrent treatment arms.

With the completion of ABTC1801, a Phase I/II Study of BGB-290 with Temozolomide in Recurrent Gliomas with IDH1/2 Mutations, a maximum tolerated dose (MTD) for adults has been found. This study will advance to evaluate preliminary efficacy using this dose in patients 13-25 years of age.

EXPLORATORY OBJECTIVES:

I. Evaluate the preliminary efficacy of BGB-290 and temozolomide in terms of progression free survival (PFS) and overall survival (OS) in Arm A and B stratified by tumor diagnosis, calculated using the Kaplan-Meier method with a goal of improving the historical high grade glioma progression free survival of 10% and overall survival of 20% at 2 years.

II. Assess the mutational landscape studies via whole-exome sequencing (WES).

III. Assessment of gene expression patterns using ribonucleic acid (RNA) sequencing (RNAseq).

IV. Assess the methylation profiling with Infinium methylation assays.

V. Assess the oncometabolite profiling via liquid chromatography (LC)/mass spectrometry (MS)-MS.

VI. Assess the intratumoral drug level assessments via LC/MS-MS.

VII. To assess Quality of Life (QOL) and cognitive measures in adolescent and young adult patients with newly diagnosed and recurrent mutant gliomas.

VIII. To assess patient and/or proxy satisfaction with study participation via patient-reported outcome (PRO) measures in the context of race ethnicity and other health related social risks.

IX. To assess on therapy toxicity in the context of race, ethnicity and other health related social risks.

OUTLINE: Participants are assigned to 1 of 2 cohorts. The dose escalation component of the trial has been completed, which included patients ages 13-17 and the study will proceed with enrolling patients ages 13-25 years old onto the expansion cohort and target validation component at the ABTC pre-determined dose.

Arm A: Newly diagnosed IDH1/2-mutant high-grade glioma patients receive PARP inhibitor BGB-290 orally (PO) twice daily (BID) on days 1-28 and temozolomide PO daily on days 1-21. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

Arm B: Recurrent IDH1/2-mutant low-grade or high-grade glioma patients receive PARP inhibitor BGB-290 orally (PO) twice daily (BID) on days 1-28 and temozolomide PO daily on days 1-21. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

COHORT B0: Recurrent IDH1/2-mutant low-grade or high-grade glioma patients receive PARP inhibitor BGB-290 PO for 7 days pre-surgery at the ABTC-determined MTD. After recovery from surgery (14-28 days), the patient will proceed to the efficacy component of the trial.

After completion of study treatment, patients are followed up for 5 years. If participants are co-enrolled on the PNOC COMP protocol, participants will be followed under the PNOC COMP protocol until death or withdrawal from study.

ELIGIBILITY:
Inclusion Criteria:

* Arm A Only: Participants must have histologically confirmed World Health Organization (WHO) grade III-IV newly diagnosed IDH1/2-mutant glioma.
* Arm B Only: WHO grades I-IV recurrent IDH1/2 mutant glioma. Participants in Arm B must have magnetic resonance imaging (MRI) confirming progressive disease; re-biopsy is encouraged, but not required at the time of recurrence for confirmation.
* Participants with a primary spinal tumor, secondary glioma, or multifocal disease in the brain, but without evidence of diffuse leptomeningeal spread, are eligible. In cases where there are questions about multifocality versus diffuse leptomeningeal spread, the study chair or co-chair must be contacted to make a final decision on eligibility.
* Participants must have IDH1 or IDH2 mutation associated with neomorphic activity of the encoded proteins.
* Participants must be willing to provide archival formalin-fixed embedded (FFPE) and frozen tissue specimens for biomarker studies if available.
* Participants in Arm A must have been treated with maximal safe resection of primary tumor followed by adjuvant radiation therapy (RT). Treatment with TMZ during radiation is allowed but not required.
* Participants in Arm B must have been treated with maximal safe resection of tumor.

  * Lower grade glioma (LGG) participants who progressed after initial surgery alone are eligible. Any number of prior therapies are allowed.
  * High grade glioma (HGG) participants enrolled on Arm B must have been treated with a minimum of maximal safe resection of primary tumor followed by adjuvant RT prior to recurrence. Any number of prior therapies are allowed.
* Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: participants must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks if nitrosourea.
* Biologic agent: participants must have recovered from any toxicity related to biologic agents and received their last dose >= 7 days prior to study registration.

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval should be discussed with the study chair.
  * For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the study chair prior to registration.
* Monoclonal antibody treatment: at least three half-lives must have elapsed prior to registration, and participants on bevacizumab must have received their last dose >= 32 days prior to study registration.
* Participants in Arm A should begin therapy with TMZ and BGB-290 after completion of radiation therapy and when all other eligibility criteria are met.
* For participants in Arm B, patients must not have received radiation therapy within 4 weeks prior to the initiation of study treatment. Post-RT, the diagnosis of true progression versus pseudo-progression can be challenging when imaging modalities are exclusively used, and thus an additional resection is encouraged if clinically indicated.
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3.
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Hemoglobin >= 9 g/dL.
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or estimated creatinine clearance >= 50 mL/min (calculated using the institutional standard method).
* Total serum bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN).
* Aspartate and alanine aminotransferase (AST and ALT) =< 3 x ULN.
* Serum albumin >= 2 g/dL.
* Participants with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled.
* Participants who have neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.
* Corticosteroids: Participants who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
* The effects of BGB-290 on the developing human fetus are unknown. For this reason and because alkylating agents (such as TMZ) are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of BGB-290 or TMZ administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participants must be able to swallow capsules.
* Participants must have the ability to undergo serial MRI scans (computerized tomography [CT] cannot substitute for MRI).
* A legal parent/guardian or patient must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.
* Karnofsky >= 50 for participants > 16 years of age and Lansky >= 50 for participants =< 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Exclusion Criteria:

* Participants who are receiving any other investigational agents at any time may not be enrolled.
* Participants who have received a PARP inhibitor previously.
* Participants with active infection requiring antibiotics at time of therapy start.
* Participants with other diagnosis of malignancy.
* Participants with clinically significant active bleeding disorder, hemoptysis, or melena =< 6 months prior to day 1.
* Participants on therapeutic anti-coagulation with heparin, warfarin, or other anticoagulants:

  * Use of low-dose aspirin and/or non-steroidal anti-inflammatory agents are allowed.
  * Use of thrombolytic to establish patency of indwelling venous catheters is allowed.
  * Prophylactic anticoagulation for venous access devices is allowed as long as institutional normalized ratio (INR) is =< 1.5 and partial thromboplastin time (aPTT) =< 1.5 x institutional ULN.
  * Use of low-molecular weight heparin is allowed.
* Participants with known disseminated leptomeningeal disease.
* Participants with diffuse intrinsic pontine glioma (DIPG) are not eligible for this study.
* Unresolved acute effects of any prior therapy of grade >= 2, except for adverse events (AEs) not constituting a safety risk by investigator judgement.
* Use =< 10 days (or =< 5 half-lives, whichever is shorter) prior to day 1 or anticipated need for food or drugs known to be strong or moderate Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or strong CYP3A inducers.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TMZ or pamiparib (BGB-290).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Female participants of childbearing potential must not be pregnant or breast-feeding. Female participants of childbearing potential must have a negative serum or urine pregnancy test within 7 days of first dose.
* Human immunodeficiency virus (HIV)-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pamiparib (BGB-290) and TMZ. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Participants with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Events occurring on or after treatment on Day 1 will be classified using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Adverse events leading to treatment discontinuation will be listed.

OTHER OUTCOMES:
Progression free survival (PFS) | Up to 5 years
  The analyses of PFS will include patients who have received any amount of study treatment. PFS is defined as the time from the first day of study treatment with until documented disease progression or death, whichever occurs first. For patients who do not have documented progressive disease (PD) or death before the end of the study or who are lost to follow-up, PFS will be censored at the day of the last clinical assessment. Data will be summarized by Kaplan-Meier method.
Overall survival (OS) | Up to 5 years
  The analyses of OS will include patients who have received any amount of study treatment. OS is defined as the time from the first dose of study treatment to the time of death from any cause on study. For patients who do not die before the end of the study or who are lost to follow-up, OS will be censored at the date of last contact. Data will be summarized by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Joseph M. Sanzari Children's Hospital at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification.
Supporting Information: Study Protocol